CLINICAL TRIAL: NCT02314156
Title: Intra-mammary Distribution of Transdermal Telapristone Versus Oral Telapristone: A Randomized Window Trial in Women Undergoing Mastectomy
Brief Title: Transdermal or Oral Telapristone Acetate in Treating Patients Undergoing Mastectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NCI 2013-01-03; NCI-2014-02412 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00035; NCI 2013-01-03 (Other: Northwestern University); NWU2013-01-03 (Other: DCP); HHSN26100003 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: BRCA1 Mutation Carrier; BRCA2 Mutation Carrier; Ductal Breast Carcinoma In Situ; Lobular Breast Carcinoma In Situ; Stage 0 Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms | interventions — telapristone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (transdermal telapristone acetate) (Experimental): Patients receive telapristone acetate transdermally and placebo PO QD for 4 weeks.
  Interventions: Drug: Telapristone Acetate; Other: Placebo; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm II (oral telapristone acetate) (Active Comparator): Patients receive placebo transdermally and telapristone acetate PO QD for 4 weeks.
  Interventions: Drug: Telapristone Acetate; Other: Placebo; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Telapristone Acetate — Given transdermally
  Other Names: CDB-4124; Proellex; Progenta
  Arms: Arm I (transdermal telapristone acetate)
Other: Placebo — Given PO
  Other Names: PLCB
  Arms: Arm I (transdermal telapristone acetate)
Drug: Telapristone Acetate — Given PO
  Other Names: CDB-4124; Proellex; Progenta
  Arms: Arm II (oral telapristone acetate)
Other: Placebo — Given transdermally
  Other Names: PLCB
  Arms: Arm II (oral telapristone acetate)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized trial studies transdermal or oral telapristone acetate in treating patients undergoing surgery to remove the breast (mastectomy). Telapristone acetate may help prevent breast cancer from forming in premenopausal women. Giving telapristone acetate transdermally may be safer and have fewer side effects than oral administration.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate that mean levels of telapristone (telapristone acetate) in breast tissue following gel application will result in levels that are not more than 50% lower than those following oral administration.

SECONDARY OBJECTIVES:

I. To assess whether plasma concentrations of telapristone are significantly lower with transdermal than oral therapy.

II. To compare within-breast variation of breast tissue concentration in transdermal and oral groups.

III. To measure changes in cell proliferation (marker of proliferation (Ki-67 labeling index).

IV. Explore changes in gene expression in breast tissue related to telapristone therapy.

V. Assess change in serum progesterone associated with telapristone therapy. VI. Assess the safety and tolerability of oral and transdermal administration. VII. Assess symptom measurements using BESS Questionnaire

OUTLINE: Participants are randomized to 1 of 2 treatment arms.

ARM I (TRANSDERMAL TELAPRISTONE ACETATE): Patients receive telapristone acetate transdermally and placebo orally (PO) once daily (QD) for 4 weeks.

ARM II (ORAL TELAPRISTONE ACETATE): Patients receive placebo transdermally and telapristone acetate PO QD for 4 weeks.

After completion of study treatment, patients are followed up at day 60.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for unilateral or bilateral mastectomy for breast cancer therapy, pathology confirmed stage 0-II (including ductal carcinoma in situ), or prophylaxis (breast cancer, early onset [BRCA] mutation carriers, women with strong family history or lobular carcinoma in situ or other conditions where prophylactic mastectomy has been elected)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Total bilirubin < 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) < 2.5 x ULN
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x ULN
* Creatinine < 2 x ULN
* Alkaline phosphatase < 2.5 x ULN
* Blood urea nitrogen < 2 x ULN
* Willing to use non-hormonal contraception (adequate barrier-type contraception or intrauterine device [IUD]) from the time the pregnancy test is performed for the duration of study participation, and 30 days after study drug cessation (for women of childbearing potential only)
* Ability to understand and the willingness to sign a written informed consent document
* Willing and able to schedule mastectomy 4 weeks (+/- 7days) following start of study agent
* Willing to avoid exposing breast skin to natural or artificial sunlight (i.e. tanning beds) for the duration of study agent dosing
* Negative urine pregnancy test result, for participants of child bearing potential, within 5 days prior to first dose of study medication; female of child-bearing potential is any woman (regardless of sexual orientation, whether she has undergone a tubal ligation, or remains celibate by choice) who meets the following criteria: has not undergone a hysterectomy or bilateral oophorectomy; OR has had a menstrual period at any time in the preceding 12 consecutive months)
* Willing to use alcohol in moderation while taking study agent

Exclusion Criteria:

* The presence of skin invasion by the breast cancer, or inflammatory changes with skin edema AND erythema. Note: Paget's disease is permitted.
* Women receiving a "nipple delay" procedure prior to mastectomy.
* Women with skin diseases (psoriasis, eczema) on breast.
* A history of thromboembolic disorder or cerebral vascular disease
* Use of oral contraceptives or other hormonal treatments within eight weeks prior to the randomization or during the period of the study; women should not have used Depo-Provera in the preceding 6 months; use of hormone coated IUD like Mirena is allowed
* Participants may not have received any other investigational agents in the previous 3 months
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to telapristone (i.e. other progesterone antagonists)
* Taken tamoxifen or other selective estrogen/progesterone receptor modulators (SERMs/SPRMs) within two years prior to entering study or been required to discontinue SERM therapy due to thromboembolic or uterine toxicity
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of prior breast cancer-specific therapy within the previous 2 years; previous unilateral radiation in women scheduled for mastectomy of the contralateral side is allowed
* Pregnant or breastfeeding
* Currently taking spironolactone
* Recent history (within 6 months) of alcoholism or drug abuse
* Known active infection with human immunodeficiency virus (HIV), hepatitis A, B, or C

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Khan, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, West Hollywood, California
  - Northwestern University, Chicago, Illinois
  - Memorial Sloan-Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Transdermal Telapristone Acetate): Participants receive telapristone acetate transdermally and placebo PO QD for 4 weeks.
  Telapristone Acetate: Given transdermally applied to both breast skin
  Placebo: Given PO
- Arm II (Oral Telapristone Acetate): Patients receive placebo transdermally and telapristone acetate PO QD for 4 weeks.
  Telapristone Acetate: Given PO
  Placebo: Given transdermally applied to both breast skin
Period: Overall Study
Arm/Group | Arm I (Transdermal Telapristone Acetate) | Arm II (Oral Telapristone Acetate)
Started | 33 | 34
Completed | 31 | 34
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Transdermal Telapristone Acetate) | Arm II (Oral Telapristone Acetate) | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (9.27) | 49.3 (13.41) | 48.6 (11.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 27 | 26 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Mean Levels of Telapristone Acetate in Breast Tissue
Description: Post-therapy mean levels of telapristone acetate in breast tissue.
Time Frame: At the time of mastectomy, up to 5 weeks from baseline
Population: Participants with post-therapy breast tissue samples
Measure: Median (Inter-Quartile Range); unit: ng/g
Arm/Group | Arm I (Transdermal Telapristone Acetate) | Arm II (Oral Telapristone Acetate)
Number analyzed (Participants) | 28 | 31
ng/g | 2.82 [1.37 to 5.47] | 103 [46.3 to 336]

2. Secondary Outcome: Plasma Concentrations of Telapristone Acetate
Description: Post-therapy plasma concentrations of telapristone acetate.
Time Frame: At the time of mastectomy, up to 5 weeks from baseline
Population: Participants with plasma samples post-therapy.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm I (Transdermal Telapristone Acetate) | Arm II (Oral Telapristone Acetate)
Number analyzed (Participants) | 28 | 32
ng/ml | 0.93 [0.39 to 1.41] | 69.0 [32.8 to 138]

3. Secondary Outcome: Within-breast Variation of Breast Tissue Concentration of Telapristone Acetate
Description: Post-therapy concentrations of telapristone acetate in 5 locations within breast tissue.
Time Frame: At the time of mastectomy, up to 5 weeks from baseline
Population: Participants with post-therapy breast tissue samples.
Measure: Median (Inter-Quartile Range); unit: ng/g
Arm/Group | Arm I (Transdermal Telapristone Acetate) | Arm II (Oral Telapristone Acetate)
Number analyzed (Participants) | 28 | 31
ng/g
  Central Subalveolar | 1.73 [1.15 to 3.61] | 63.7 [37.7 to 205]
  Central Deepest | 5.09 [2.12 to 10.8] | 133 [34.9 to 248]
  Lateral Surface | 6.76 [2.55 to 15.5] | 214 [104 to 354]
  Lateral Center | 2.42 [0.42 to 5.2] | 85.5 [40.6 to 292]
  Medial Center | 2.79 [1.44 to 4.27] | 121 [37.9 to 389]

4. Secondary Outcome: Changes in Cell Proliferation
Description: Changes in cell proliferation (Ki67 labeling index) measured in percentage of positive cells from baseline to mastectomy by tumor status in ER positive tumors.
Time Frame: Baseline to mastectomy (up to 5 weeks)
Population: Participants with ER positive tumors.
Measure: Median (Inter-Quartile Range); unit: % positive
Arm/Group | Arm I (Transdermal Telapristone Acetate) | Arm II (Oral Telapristone Acetate)
Number analyzed (Participants) | 17 | 15
% positive | -0.67 [-2.8 to 0.57] | 5.2 [-5.9 to 6.9]

5. Secondary Outcome: Changes in Serum Sex Hormone Concentrations: Estradiol
Description: Change in estradiol in premenopausal women from baseline to post-intervention compared between treatment groups
Time Frame: Baseline to mastectomy, up to 5 weeks post-intervention
Population: Premenopausal women
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm I (Transdermal Telapristone Acetate) | Arm II (Oral Telapristone Acetate)
Number analyzed (Participants) | 18 | 18
pg/ml | 95.9 [75.1 to 135] | -23.7 [-97.5 to -1.70]

6. Secondary Outcome: Change in Symptoms as Captured in the Breast Cancer Prevention Trial (BCPT) Eight Symptom Scale (BESS) Questionnaire
Description: Mean change in symptoms as captured using the Breast Cancer Prevention Trial (BCPT) Eight Symptom Scale (BESS) questionnaire. A patient reported outcome, scores range from 0 (Not at All) to 4 (Extremely) when asked about experiencing symptoms. A positive change in scores indicates an increase in symptoms experienced and a negative change in scores indicates a decrease in symptoms experienced
Time Frame: Baseline to mastectomy (up to 5 weeks)
Population: participants
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Transdermal Telapristone Acetate) | Arm II (Oral Telapristone Acetate)
Number analyzed (Participants) | 31 | 32
score on a scale
  Cognitive | -0.61 (0.53) | -0.88 (0.43)
  Body Pain | -0.81 (0.44) | -0.78 (0.43)
  Vasomotor | 0.71 (0.26) | 0.09 (0.23)
  Gastrointestinal | 0.16 (0.35) | -0.34 (0.11)
  Sexual problems | -0.29 (0.24) | -0.28 (0.19)
  Bladder | -0.32 (0.18) | -0.38 (0.18)
  Body Image | 0.52 (0.34) | -0.16 (0.25)
  Vaginal | -0.35 (0.20) | 0.19 (0.27)

7. Secondary Outcome: Changes in Serum Sex Hormone Concentrations: Progesterone
Description: Change in progesterone in premenopausal women from baseline to post-intervention compared between treatment groups
Time Frame: Baseline to mastectomy (up to 5 weeks)
Population: Premenopausal women
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm I (Transdermal Telapristone Acetate) | Arm II (Oral Telapristone Acetate)
Number analyzed (Participants) | 18 | 18
ng/ml | 0.19 [-0.12 to 1.51] | -2.36 [-10.1 to 0]

8. Secondary Outcome: Changes in Serum Sex Hormone Concentrations: FSH
Description: Change in FSH in premenopausal women from baseline to post-intervention compared between treatment groups
Time Frame: Baseline to mastectomy (up to 5 weeks)
Population: Premenopausal women
Measure: Median (Inter-Quartile Range); unit: mIU
Arm/Group | Arm I (Transdermal Telapristone Acetate) | Arm II (Oral Telapristone Acetate)
Number analyzed (Participants) | 18 | 18
mIU | 1.91 [-0.40 to 4.28] | 0.30 [-2.84 to 2.21]

ADVERSE EVENTS:
Time Frame: AEs collected from the time informed consent was signed and baseline procedures were completed through up to 5 weeks post-intervention.
Arm/Group | Arm I (Transdermal Telapristone Acetate) | Arm II (Oral Telapristone Acetate)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 25/33 | 21/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Transdermal Telapristone Acetate) (N=33) | Arm II (Oral Telapristone Acetate) (N=34)
General disorders and administrative site condition - other specify (General disorders) | 6 (10) | 7 (10) — application site reaction
Headache (Nervous system disorders) | 5 (5) | 7 (15)
Hot flashes (Vascular disorders) | 13 (23) | 7 (10)
Nausea (Gastrointestinal disorders) | 6 (7) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT02314156/Prot_SAP_ICF_000.pdf